CLINICAL TRIAL: NCT03893825
Title: A Study to Evaluate the Safety, Tolerability, and Effect of Risperidone Extended-Release Injectable Suspension (TV-46000) for Subcutaneous Use as Maintenance Treatment in Adult and Adolescent Patients With Schizophrenia
Brief Title: A Study to Test if TV-46000 is Safe for Maintenance Treatment of Schizophrenia
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV46000-CNS-30078; 2019-000063-24 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TV-46000 q1m (Experimental): Participants will receive a subcutaneous (SC) injection of TV-46000 at baseline and every 4 weeks (q4w) thereafter for up to 56 weeks. The maximal dose administered to adult participants is comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents is comparable to 4 mg/day.
  Interventions: Drug: TV-46000
- TV-46000 q2m (Experimental): Participants will receive an SC injection of TV-46000 at baseline and every 8 weeks (q8w) thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter for up to 56 weeks. The maximal dose administered to adult participants is comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents is comparable to 4 mg/day.
  Interventions: Drug: TV-46000; Drug: Placebo

INTERVENTIONS:
Drug: TV-46000 — TV-46000 will be administered per dose and schedule specified in the arm description.
  Other Names: Risperidone
Drug: Placebo — Placebo matching to TV-46000 will be administered per schedule specified in the arm description.
  Arms: TV-46000 q2m

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of TV-46000. The primary safety and tolerability endpoint is the frequency of all adverse events, including serious adverse events. For new participants, the total duration of participant participation in the study is planned to be up to 80 weeks (including a screening period of up to 4 weeks, a 12-week oral conversion/stabilization stage [Stage 1], a 56-week double-blind maintenance stage [Stage 2], and a follow-up period [8 weeks]). For roll-over participants, the total duration of participant participation in the study is planned to be up to 64 weeks (including up to 56 weeks in the maintenance stage [Stage 2] and a follow-up period [8 weeks]). Participants who started Stage 2 who relapse or meet 1 or more of the withdrawal criteria should be invited to perform the Early Termination visit as soon as possible within 4 weeks of the last injection. Participants who withdraw from the study before completing the 56-week maintenance stage will have follow-up procedures and assessments performed at their follow-up visits. During the follow-up period, participants will be treated according to the investigator's judgment.

All participants will be treated with active drug.

ELIGIBILITY:
Inclusion Criteria:

Participants Rolling Over from the Pivotal Efficacy Study TV46000-CNS-30072:

* The participant must have participated in the pivotal efficacy study (Study TV46000-CNS-30072) without experiencing relapse events and without important protocol deviations.
* If the participant was taking antidepressants or mood stabilizers in Study TV46000-CNS-30072, no dose changes or initiation of treatment with these medications will be permitted.
* The participant, in the investigator's judgment, requires chronic treatment with an antipsychotic medication.
* The participant is able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens (oral and SC administration) and non-use of prohibited concomitant medications; can read and understand the written word in order to complete participant-reported outcomes measures; and can be reliably rated on assessment scales.
* The participant has had a stable place of residence for the previous 3 months before the baseline visit in this study, and changes in residence are not anticipated over the course of study participation.
* The participant has no significant life events (such as pending loss of housing, family status change, long travel abroad, surgery, etc) that could affect study outcomes expected throughout the period of study participation.
* Women of childbearing potential and sexually active female adolescents must agree not to try to become pregnant, and, unless they have exclusively same-sex partners, must agree to use a highly effective method of contraception and agree to continue use of this method beginning 1 month before the first administration of study drug and for the duration of the study and for 120 days after the last injection of study drug.
* The participant, if adult or adolescent male, is surgically sterile, or, if capable of producing offspring, has exclusively same-sex partners or is currently using an approved method of birth control and agrees to the continued use of this method for the duration of the study (and for 120 days after the last dose of study drug). Male participants with sex partners who are women of childbearing potential must use condoms even if surgically sterile. In addition, male participants may not donate sperm for the duration of the study and for 120 days after taking the study drug.

New Participants (Not Rolling Over from the Pivotal Efficacy Study TV46000-CNS-30072):

* The participant has a diagnosis of schizophrenia
* The participant has been responsive to an antipsychotic treatment (other than clozapine) in the past year based on investigator judgment (and discussions with family members, caregivers, or healthcare professionals as applicable).
* The participant, in the investigator's judgment, requires chronic treatment with an antipsychotic medication.
* The participant is able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens (oral and sc administration) and non-use of prohibited concomitant medications; can read and understand the written word in order to complete participant-reported outcomes measures; and can be reliably rated on assessment scales.
* The participant has had a stable place of residence for the previous 3 months before screening, and changes in residence are not anticipated over the course of study participation.
* The participant has no significant life events (such as pending loss of housing, family status change, long travel abroad, surgery, etc) that could affect study outcomes expected throughout the period of study participation.
* The participant has a body mass index between 18.0 and 38.0 kilograms (kg)/square meter (m^2), inclusive.
* Women of childbearing potential and sexually active female adolescents must agree not to try to become pregnant, and, unless they have exclusively same-sex partners, must agree to use a highly effective method of contraception and agree to continue use of this method beginning 1 month before the first administration of study drug and for the duration of the study and for 120 days after the last injection of study drug.
* The participant, if adult or adolescent male, is surgically sterile, or, if capable of producing offspring, has exclusively same-sex partners or is currently using an approved method of birth control and agrees to the continued use of this method for the duration of the study (and for 120 days after the last dose of study drug). Male participants with sex partners who are women of childbearing potential must use condoms even if surgically sterile. In addition, male participants may not donate sperm for the duration of the study and for 120 days after taking the study drug.
* Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

Participants Rolling Over from the Pivotal Efficacy Study TV46000-CNS-30072:

* The participant has a finding in the baseline 12-lead electrocardiogram (ECG) that is considered clinically significant in the judgment of the investigator.
* Poor compliance with study procedures (in the opinion of the investigator or sponsor) during the pivotal efficacy Study TV46000-CNS-30072. This should be discussed on a case-by-case basis.

New Participants (Not Rolling Over from the Pivotal Efficacy Study TV46000-CNS-30072) and Roll-Over Participants:

* The participant is currently on clozapine or has received electroconvulsive therapy in the last 12 months.
* The participant has a history of epilepsy or seizures, neuroleptic malignant syndrome, tardive dyskinesia, or other medical condition that would expose the participant to undue risk.
* The participant has a positive serology for human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B surface antigen, and/or hepatitis C.
* The participant has current or a history of known hypersensitivity to risperidone or any of the excipients of TV-46000 or the oral formulation of risperidone used in the stabilization phase.
* The participant has a substance use disorder, including alcohol and benzodiazepines but excluding nicotine and caffeine.
* The participant is a pregnant or lactating female.
* The participant has used an investigational drug other than TV-46000 within 3 months prior to screening or has participated in a non-drug clinical trial within 30 days prior to screening.
* Vulnerable participants (for example, people kept in detention).
* Additional criteria apply, please contact the investigator for more information.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (90):
- United States (67):
  - Teva Investigational Site 14391, Phoenix, Arizona
  - Teva Investigational Site 14401, Scottsdale, Arizona
  - Teva Investigational Site 14405, Tucson, Arizona
  - Teva Investigational Site 14796, Rogers, Arkansas
  - Teva Investigational Site 14811, Anaheim, California
  - Teva Investigational Site 14794, Bellflower, California
  - Teva Investigational Site 14776, Colton, California
  - Teva Investigational Site 14802, Costa Mesa, California
  - Teva Investigational Site 14773, Culver City, California
  - Teva Investigational Site 14774, Glendale, California
  - Teva Investigational Site 14817, La Habra, California
  - Teva Investigational Site 14771, Lemon Grove, California
  - Teva Investigational Site 14863, Long Beach, California
  - Teva Investigational Site 14816, Montclair, California
  - Teva Investigational Site 14786, Oakland, California
  - Teva Investigational Site 14827, Oceanside, California
  - Teva Investigational Site 14777, Orange, California
  - Teva Investigational Site 14815, Pico Rivera, California
  - Teva Investigational Site 14785, San Bernardino, California
  - Teva Investigational Site 14818, San Diego, California
  - Teva Investigational Site 14788, Torrance, California
  - Teva Investigational Site 14783, Coral Gables, Florida
  - Teva Investigational Site 14865, Hialeah, Florida
  - Teva Investigational Site 14787, Hialeah, Florida
  - Teva Investigational Site 14814, Hialeah, Florida
  - Teva Investigational Site 14861, Homestead, Florida
  - Teva Investigational Site 14390, Lake Mary, Florida
  - Teva Investigational Site 14799, Lauderhill, Florida
  - Teva Investigational Site 14389, Maitland, Florida
  - Teva Investigational Site 14875, Miami, Florida
  - Teva Investigational Site 14400, Miami, Florida
  - Teva Investigational Site 14832, Miami, Florida
  - Teva Investigational Site 14810, North Miami, Florida
  - Teva Investigational Site 14860, Tampa, Florida
  - Teva Investigational Site 14396, West Miami, Florida
  - Teva Investigational Site 14821, Decatur, Georgia
  - Teva Investigational Site 14770, Marietta, Georgia
  - Teva Investigational Site 14415, Norcross, Georgia
  - Teva Investigational Site 14829, Chicago, Illinois
  - Teva Investigational Site 14805, Hoffman Estates, Illinois
  - Teva Investigational Site 14871, Lincolnwood, Illinois
  - Teva Investigational Site 14862, Lake Charles, Louisiana
  - Teva Investigational Site 14869, Monroe, Louisiana
  - Teva Investigational Site 14866, Gaithersburg, Maryland
  - Teva Investigational Site 14764, Glen Burnie, Maryland
  - Teva Investigational Site 14791, St Louis, Missouri
  - Teva Investigational Site 14813, St Louis, Missouri
  - Teva Investigational Site 14826, St Louis, Missouri
  - Teva Investigational Site 14809, Las Vegas, Nevada
  - Teva Investigational Site 14414, Las Vegas, Nevada
  - Teva Investigational Site 14792, Berlin, New Jersey
  - Teva Investigational Site 14772, Cedarhurst, New York
  - Teva Investigational Site 14876, New York, New York
  - Teva Investigational Site 14780, Staten Island, New York
  - Teva Investigational Site 14867, Hickory, North Carolina
  - Teva Investigational Site 14416, Beachwood, Ohio
  - Teva Investigational Site 14763, Cincinnati, Ohio
  - Teva Investigational Site 14782, Dayton, Ohio
  - Teva Investigational Site 14859, Garfield Heights, Ohio
  - Teva Investigational Site 14793, Media, Pennsylvania
  - Teva Investigational Site 14778, Charleston, South Carolina
  - Teva Investigational Site 14868, Memphis, Tennessee
  - Teva Investigational Site 14801, Houston, Texas
  - Teva Investigational Site 14807, Irving, Texas
  - Teva Investigational Site 14393, Plano, Texas
  - Teva Investigational Site 14856, Richardson, Texas
  - Teva Investigational Site 14395, Bellevue, Washington
- Bulgaria (8):
  - Teva Investigational Site 59148, Burgas
  - Teva Investigational Site 59152, Kazanlak
  - Teva Investigational Site 59151, Lovech
  - Teva Investigational Site 59149, Novi Iskar
  - Teva Investigational Site 59144, Sofia
  - Teva Investigational Site 59154, Varna
  - Teva Investigational Site 59150, Varna
  - Teva Investigational Site 59146, Vratsa
- Canada (5):
  - Teva Investigational Site 11169, Edmonton, Alberta
  - Teva Investigational Site 11171, Calgary, AL
  - Teva Investigational Site 11173, Vancouver, British Columbia
  - Teva Investigational Site 11170, Chatham, Ontario
  - Teva Investigational Site 11174, Montreal, Quebec
- France (4):
  - Teva Investigational Site 35259, Clermont-Ferrand
  - Teva Investigational Site 35257, Douai
  - Teva Investigational Site 35260, Nice
  - Teva Investigational Site 35256, Toulon
- Israel (6):
  - Teva Investigational Site 80162, Afula
  - Teva Investigational Site 80161, Ashkelon
  - Teva Investigational Site 80156, Haifa
  - Teva Investigational Site 80155, Hod HaSharon
  - Teva Investigational Site 80157, Ramat Gan
  - Teva Investigational Site 80160, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request

REFERENCES:
- [Derived] Kane JM, Tohami O, Franzenburg KR, Suett M, Sharon N, Merenlender-Wagner A, Eshet R, Harary E, Correll CU. Effects of Long-Term Treatment with TV-46000 on Symptom Improvement Over Time in Stabilized Patients with Schizophrenia. CNS Drugs. 2025 Nov 21. doi: 10.1007/s40263-025-01240-1. Online ahead of print. PMID 41272239
- [Derived] Correll CU, Knebel H, Harary E, Eshet R, Tohami O, Suett M, Sharon N, Franzenburg KR, Kane JM. Safety Outcomes with the Long-Acting Subcutaneous Antipsychotic TV-46000 in Schizophrenia: A Post Hoc Analysis of Behavioral, Neuromotor, Endocrine, and Cardiometabolic Outcomes from Two Phase 3 Studies. CNS Drugs. 2025 Nov;39(11):1139-1156. doi: 10.1007/s40263-025-01197-1. Epub 2025 Jul 29. PMID 40730715
- [Derived] Kane JM, Eshet R, Harary E, Tohami O, Elgart A, Knebel H, Sharon N, Suett M, Franzenburg KR, Davis GL 3rd, Correll CU. A Long-Term Safety and Tolerability Study of TV-46000 for Subcutaneous Use in Patients with Schizophrenia: A Phase 3, Randomized, Double-Blinded Clinical Trial. CNS Drugs. 2024 Aug;38(8):625-636. doi: 10.1007/s40263-024-01102-2. Epub 2024 Jul 2. PMID 38954317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who did not experience a relapse and completed Study TV46000-CNS-30072 (NCT03503318) (roll-over participants) and new participants entered this study. Open-label oral risperidone (at a dose of 2 to 5 milligrams [mg]/day, based on clinical judgment) for 12 weeks was given to stabilize new participants to the treatments before randomization.
Pre-assignment Details: Participants who were treated with TV-46000 once monthly (q1m) or once every 2 months (q2m) during Study TV46000-CNS-30072, continued their assigned treatment. Participants who were treated with placebo during Study TV46000-CNS-30072 were randomized in 1:1 to receive TV-46000 q1m or q2m subcutaneous (SC) injections at equivalent to oral dose on which they were stabilized.
Groups:
- TV-46000 q1m: Participants received an SC injection of TV-46000 at baseline and every 4 weeks (q4w) thereafter for up to 56 weeks. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day.
- TV-46000 q2m: Participants received an SC injection of TV-46000 at baseline and every 8 weeks (q8w) thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter for up to 56 weeks. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day.
Period: Overall Study
Arm/Group | TV-46000 q1m | TV-46000 q2m
Started | 174 | 162
Received at Least 1 Dose of Study Drug | 172 | 162
Completed | 135 | 122
Not Completed | 39 | 40
Not completed — Death | 2 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 19 | 21
Not completed — Protocol deviation | 1 | 0
Not completed — Lost to Follow-up | 10 | 10
Not completed — Other than specified | 7 | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants who were randomized either in Study TV46000-CNS-30072 for roll-over participants or in Study TV46000-CNS-30078.
Groups:
- TV-46000 q1m: Participants received an SC injection of TV-46000 at baseline and q4w thereafter for up to 56 weeks. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day.
- TV-46000 q2m: Participants received an SC injection of TV-46000 at baseline and q8w thereafter, and a placebo SC injection 4 weeks after baseline and q8w thereafter for up to 56 weeks. The maximal dose administered to adult participants was comparable to an oral risperidone dose of 5 mg/day, and the maximal dose administered to adolescents was comparable to 4 mg/day.
- Total: Total of all reporting groups
Arm/Group | TV-46000 q1m | TV-46000 q2m | Total
Number analyzed (Participants) | 174 | 162 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.28) | 49.8 (11.51) | 50.6 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 120
  Male | 113 | 103 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 51 | 107
  Not Hispanic or Latino | 118 | 110 | 228
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 80 | 67 | 147
  Race: Black or African American | 91 | 90 | 181
  Race: Asian | 1 | 2 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Not reported | 1 | 1 | 2
  Race: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 64
Population: The safety analysis set included all participants who received at least 1 dose of TV46000 in TV-46000-CNS-30072 study or in TV46000-CNS-30078 study.
Measure: Count of Participants; unit: Participants
Arm/Group | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 172 | 162
Participants | 64 | 74

2. Other Pre Specified Outcome: Number of Participants Who Were Withdrawn From the Treatment
Description: The number of participants who were withdrawn from the treatment due to any reason has been reported. The safety analysis set included all participants who received at least 1 dose of TV46000 in TV-46000-CNS-30072 study or in TV46000-CNS-30078 study.
Time Frame: Baseline up to Week 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 172 | 162
Participants
  Death | 2 | 1
  Adverse event | 2 | 5
  Withdrawal by participant | 21 | 25
  Non-compliance with study drug | 1 | 0
  Protocol deviation | 2 | 1
  Lost-to-follow up | 5 | 7
  Lack of efficacy | 1 | 0
  Relapse | 3 | 3
  Other | 11 | 11

3. Primary Outcome: Number of Participants With SAEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section. The safety analysis set included all participants who received at least 1 dose of TV46000 in TV-46000-CNS-30072 study or in TV46000-CNS-30078 study.
Time Frame: Baseline up to Week 64
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TV-46000 q1m | TV-46000 q2m
Number analyzed (Participants) | 172 | 162
Participants | 8 | 11

ADVERSE EVENTS:
Time Frame: Baseline up to Week 64
Description: The safety analysis set included all participants who received at least 1 dose of TV46000 in TV-46000-CNS-30072 study or in TV46000-CNS-30078 study. No study drug was administered during the open-label stabilization period. All treatment-emergent adverse events are presented.
Arm/Group | TV-46000 q1m | TV-46000 q2m
All-Cause Mortality (participants affected / at risk) | 2/172 | 1/162
Serious Adverse Events (participants affected / at risk) | 8/172 | 11/162
Other Adverse Events (participants affected / at risk) | 10/172 | 12/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-46000 q1m (N=172) | TV-46000 q2m (N=162)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-46000 q1m (N=172) | TV-46000 q2m (N=162)
Injection site nodule (General disorders) | 3 (6) | 9 (13)
Injection site pain (General disorders) | 9 (24) | 7 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT03893825/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03893825/SAP_001.pdf